CLINICAL TRIAL: NCT04152369
Title: "Comparison of the Effectiveness of 24-hour and 72-hour Peri-procedural Antimicrobial Prophylaxis in Patients Undergoing Endourological Procedures and ESWL Presenting With Asymptomatic Bacteriuria of Enterobacteriacae ESBL+ Origin"
Brief Title: "Peri-operative Antimicrobial Prophylaxis in Patients With Asymptomatic Bacteriuria of Enterobacteriacae ESBL+ Origin"
Acronym: ESBL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Principal Investigator, Marcin Radko, Principal Investigator, Military Institute od Medicine National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0000000495
Record Dates: First submitted 2019-10-29; First posted 2019-11-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Antimicrobial Prophylaxis; Asymptomatic Bacteriuria
Keywords: ESBL+; Antimicrobial prophylaxis
MeSH Terms: interventions — Lithotripsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24 hour prophylaxis (Active Comparator): In this group patients received a AMP for the day of the procedure
  Interventions: Procedure: Anti-microbial prophylaxis for an endourological procedure or ESWL
- 72 hour prophylaxis (Active Comparator): In this group patients received a AMP one day prior, on the day of the procedure and the following day.
  Interventions: Procedure: Anti-microbial prophylaxis for an endourological procedure or ESWL

INTERVENTIONS:
Procedure: Anti-microbial prophylaxis for an endourological procedure or ESWL — anti-microbial prophylaxis according to urine culture results

SUMMARY:
The aim of the study is to determine optimal safe duration of antibiotic prophylaxis in patients undergoing endourological procedures and ESWL, presenting with asymptomatic bacteriuria caused by multi-drug resistant bacterial strains. In this study we compare safety and efficacy of a one-day vs. three-day AMP (Antimicrobial Prophylaxis) in the above mentioned group of patients.

DETAILED DESCRIPTION:
Patients with positive urine culture with Enterobacteriacae ESBL + resistance mechanism upon admission for endourological procedure or ESWL were subjected to body temperature measurement and laboratory tests: smear from the anus towards the presence of alarm pathogens, urinalysis, control urine culture, blood count, CRP (C-reactive protein), procalcitonin (PCT). After confirming the occurrence of asymptomatic bacteriuria, the patients were randomized to two groups - a one-day and three-day period lasting perioperative antibiotic prophylaxis. In both groups on the following day after the procedure (24 hours after the procedure) and after 7 days after the procedure, laboratory tests and body temperature measurements were performed.

ELIGIBILITY:
Inclusion Criteria:

* ESBL+ asymptomatic bacteriuria
* assigned for endourological procedure
* normal CRP, PCT and WBC
* patient's consent

Exclusion Criteria:

* urinary tract infection
* raised levels of CRP, PCT, WBC
* fever
* non ESBL+ bacteriuria
* inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-07-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures and ESWL (Extracorporeal Shock Wave Lithotripsy). | 7 days
  To determine if a 1-day perioperative antibiotic prophylaxis is as safe and effective as 3-day perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures. This conclusion will be based on measurements of CRP [mg/dl] as follows: one day prior to procedure, one day post and 7 days after the procedure. The data will be statistically analyzed.
Safety and efficacy of perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures and ESWL (Extracorporeal Shock Wave Lithotripsy). | 7 days
  To determine if a 1-day perioperative antibiotic prophylaxis is as safe and effective as 3-day perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures. This conclusion will be based on measurements of WBC level [x 10^9/l] as follows: one day prior to procedure, one day post and 7 days after the procedure. The data will be statistically analyzed.
Safety and efficacy of perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures and ESWL (Extracorporeal Shock Wave Lithotripsy). | 7 days
  To determine if a 1-day perioperative antibiotic prophylaxis is as safe and effective as 3-day perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures. This conclusion will be based on measurements of levels of prokalcytonin [ng/ml] as follows: one day prior to procedure, one day post and 7 days after the procedure. The data will be statistically analyzed.
Safety and efficacy of perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures and ESWL (Extracorporeal Shock Wave Lithotripsy). | 7 days
  To determine if a 1-day perioperative antibiotic prophylaxis is as safe and effective as 3-day perioperative antibiotic prophylaxis in patients with Enterobacteriacae ESBL+ urinary tract colonization undergoing endourological procedures. This conclusion will be based on measurements of body temperature [Celsius] as follows: one day prior to procedure, one day post and 7 days after the procedure. The data will be statistically analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin A Radko, MD, Principal Investigator — Military Institute of Medicine; Henryk Zieliński, Professor, Study Chair — Military Institute of Medicine
Locations (1):
- Military Institue of Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No